CLINICAL TRIAL: NCT05340855
Title: Facebook Intervention for Preventing Opioid Relapse Among American Indian Women: Wiidookaage'Win Pilot Preparatory Study (Aim 1)
Brief Title: A Pilot Study Using Facebook to Support Opioid Recovery Among American Indian Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Christi Patten, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-000477; UG1DA040316-07S3 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Opioid Use
Keywords: American Indian; Alaska Native; Community Based Participatory Research

STUDY DESIGN:
Intervention Model Description: All study participants in Phase 3 beta test will be in the same Facebook group intervention and will view the same content.
Masking Description: This is a single arm study where every participant in Phase 3 will receive the same single intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Facebook Intervention (Experimental): In Phase 3, all participants will receive the same intervention.
  Interventions: Behavioral: Wiidookaage'win Facebook Group

INTERVENTIONS:
Behavioral: Wiidookaage'win Facebook Group — A 30-day Facebook group prototype that is moderated by two women who will post various forms of media addressing opioid recovery, mindfulness, stress management, and resiliency.

SUMMARY:
The purpose of this study is to develop a culturally relevant Facebook intervention for American Indian and Alaska Native (AIAN) women in Minnesota recovering from illicit opioid use.

DETAILED DESCRIPTION:
This one-year, Phase I, pilot preparatory study aims to develop a culturally relevant Facebook intervention for American Indian and Alaska Native (AIAN) women in Minnesota recovering from illicit opioid use. The study will consist of three phases: (1) qualitative interviews, (2) intervention content refinement and a moderator exchange (i.e., bi-directional sharing of knowledge between intervention moderators and trainers), and (3) a beta-testing period. A study-specific Community Advisory Committee (CAC) was formed whose members contributed to the study protocol and will continue to provide guidance and input on the study implementation and dissemination. At the advice of the CAC, a Native Elder woman named the study. Wiidookaage'win is an Ojibwe word that means "the place for help and time for helping," and reflects healing and community. The investigators expect the participatory approach to treatment development will result in a social media intervention with cultural relevance for Native women to maintain recovery from opioid use.

ELIGIBILITY:
Inclusion Criteria - Phase 1:

AIAN Women:

* AIAN based on self-reported race.
* Gender identity as a woman.
* Resides in Minnesota.
* At least 18 years of age age with no upper age limit.
* OUD based on the DSM-5 Checklist (American Psychiatric Association, 2013).
* Self-reports at least one month of opioid abstinence based on Timeline Follow-Back (TLFB) interview.
* Currently receiving MOUD.
* Is comfortable speaking and reading English.
* Is familiar with Facebook.
* Has access to broadband internet on a mobile phone/computer/tablet at any location.

AI/AN Health Care Providers and Stakeholders

* Health care provider or AIAN community stakeholder.
* Knowledge of Native culture and/or OUD treatment and recovery among AIAN people.
* Is comfortable speaking and reading English.
* Is familiar with Facebook.
* Has access to broadband internet on a mobile phone/computer/tablet at any location.

Having some familiarity with the Facebook platform is needed to provide feedback on content for a Facebook intervention. Access to the internet is needed to view online moderator postings for providing feedback during the interview.

Inclusion Criteria - Phase 3:

* AIAN person based on self-reported race/ethnicity.
* Gender identity as a woman.
* At least 18 years of age.
* Resides in Minnesota.
* OUD based on the DSM-5 Checklist (American Psychiatric Association, 2013).
* Self-reports at least one month of abstinence from opioid use based on TLFB interview and negative urine opiate screen.
* Currently receiving MOUD.
* Is comfortable speaking and reading English.
* Has an existing Facebook account or willing to set one up.
* Is willing and able to participate in the Facebook intervention for one month.
* Has access to broadband internet on a mobile phone/computer/tablet at any location.
* Is willing and able to travel to a community clinic in Minneapolis, Minnesota for the UDS.

Exclusion Criteria:

AIAN potential participants in Phases 1 and 3 meeting any of the exclusion criteria listed below will be excluded from study participation. Community stakeholder participants in - Phase 1 will only fail the screening if they meet the second exclusion criterion:

* Self-reports current suicidality.
* Inability or unwillingness of participant to provide verbal consent (Phase 1) or written informed consent (Phase 3).
* (Phase 3 only) Was a participant in Phase 1.

Pregnant women, lactating women, or women who plan to become pregnant will not be excluded because the treatment being evaluated is a behavioral intervention and does not involve medication or risk to the fetus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The AI/AN participants can be either transgender or cisgender women.
Enrollment: 10 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christi Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Background] Young A, Sinicrope P, Kelpin S, Roche AI, Sabaque C, Pham C, Marsch LA, Campbell ANC, Venner K, Bastian E, Nord T, Mason G, Baker L, Wyatt T, Fish A, Bart G, Patten CA. Wiidookaage'Win: A Community-Based Qualitative Approach to Developing a Facebook Group Intervention for Native Women to Support Recovery From Opioid Use. Am J Health Promot. 2024 Feb;38(2):205-218. doi: 10.1177/08901171231205355. Epub 2023 Nov 13. PMID 37955409
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Facebook Intervention: Subjects were emailed an invite link for the Facebook Intervention.
  Wiidookaage'win Facebook Group: A 30-day Facebook group prototype that was moderated by two women who posted various forms of media addressing opioid recovery, mindfulness, stress management, and resiliency.
Period: Overall Study
Arm/Group | Facebook Intervention
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Facebook Intervention
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: The Feasibility of Developing a Culturally Relevant Facebook Intervention
Description: The number of times participants engaged with the Facebook page. Define by the total times of viewing, reacting, posting, commenting and voting on any Facebook post for all participants.
Time Frame: 30 days
Measure: Median (Full Range); unit: engagement events
Arm/Group | Facebook Intervention
Number analyzed (Participants) | 10
engagement events | 33.0 [12.0 to 98.0]

2. Secondary Outcome: The Feasibility of Using Facebook as an Opioid Intervention Platform
Description: The number of participants who completed all study activities from baseline to end of study.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Facebook Intervention
Number analyzed (Participants) | 10
Participants | 9

3. Secondary Outcome: Treatment Satisfaction
Description: Treatment Satisfaction was measured using a 5-point Likert scale (1 = Strongly disagree, 5 = Strongly agree). Total scores range from 1 -5. Higher scores indicate greater satisfaction and lower scores indicate lower satisfaction.
Time Frame: 30 days
Population: One subject did not complete the post-intervention survey..
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Facebook Intervention
Number analyzed (Participants) | 9
score on a scale | 4.84 (0.18)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately 30 days
Arm/Group | Facebook Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT05340855/Prot_SAP_001.pdf
  • Informed Consent Form (2023-01-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT05340855/ICF_000.pdf